CLINICAL TRIAL: NCT06965569
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study of ALA-3000, Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy in Subjects With Treatment-Resistant Depression (TRD)
Brief Title: Multiple Ascending Dose Phase 1 Study of ALA-3000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alar Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1-23-P01
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Escitalopram; Sertraline; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects received two subcutaneous injections of "low-dose" ALA-3000 or matching volume of Placebo on Day 1 and Day 8. During the treatment period, all subjects will receive a newly initiated open-label oral antidepressants daily.
  Interventions: Drug: ALA-3000; Drug: Placebo; Drug: escitalopram, sertraline, duloxetine or venlafaxine XR
- Cohort 2 (Experimental): Subjects received two subcutaneous injections of "high-dose" ALA-3000 or matching volume of Placebo on Day 1 and Day 8. During the treatment period, all subjects will receive a newly initiated open-label oral antidepressants daily.
  Interventions: Drug: ALA-3000; Drug: Placebo; Drug: escitalopram, sertraline, duloxetine or venlafaxine XR

INTERVENTIONS:
Drug: ALA-3000 — Subcutaneous injection
Drug: Placebo — Subcutaneous injection
Drug: escitalopram, sertraline, duloxetine or venlafaxine XR — Newly initiated oral AD selected from SSRI (escitalopram or sertraline) or SNRI (duloxetine or venlafaxine XR) will be given daily

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-dose study of ALA-3000 designed to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy in subjects with treatment-resistant depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged between 18 and 65 at screening visit and is able to provide informed consent prior to initiation of any study related procedures.
2. At screening visit, subjects meet Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) criteria for single-episode major depressive disorder (MDD) or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI).
3. Subject is medically stable on basis of physical examination, medical history, vital signs (blood pressure, pulse rate, respiration rate, blood oxygen saturation, and temperature), clinical laboratory tests, and 12-lead ECG performed at screening visit, and/or prior to SC administration on Day 1. Subjects with abnormalities that are judged to be not clinically significant (NCS) at the discretion of the investigator may be included. This determination must be recorded in the subject's source documents and initialed by the investigator.
4. At screening visit, subjects must have insufficient response to at least 2 oral AD treatments, at least one of which is in the current episode of depression. Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ) will be used to assess AD treatment response during the current episode; prior medication history (e.g., medical/pharmacy/prescription records or a letter from a treating physician, etc.) will be used to determine AD treatment response in prior episode(s). If the subject's current episode of depression is > 2 years, the upper limit of duration for assessing treatment response is applicable to only the last 2 years.
5. Subject has a MADRS total score of ≥ 22 at screening.
6. Male and female subjects of childbearing potential must be willing to use a reliable method of contraception (e.g., total abstinence, condom and spermicide, intrauterine device [IUD], oral contraception which has been stable for 30 days) during the entire trial and at least 4 months after stopping the investigational product.
7. Female subjects of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) at screening visit and a negative urine pregnancy test prior to SC administration on Day 1.
8. Male and female subjects must agree not to donate sperm or eggs (ova, oocytes) during the study and for at least 3 months after receiving the investigational drug.
9. Agree to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Subject has a history of, or current signs and symptoms of, liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, metabolic disturbances, or fibromyalgia.
2. Subject has uncontrolled hypertension despite diet, exercise or a stable dose of a permitted anti-hypertensive treatment at screening visit, or prior to SC administration on Day 1 (defined as a supine SBP > 140 mmHg or DBP > 90 mmHg); or any past history of hypertensive crisis.
3. Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 × the upper limit of normal (ULN) or total bilirubin > 1.5 × ULN.
4. Subjects with history of or current DSM-5 diagnosis of psychotic disorder, or MDD with psychotic features, post-traumatic stress disorder (PTSD), bipolar or related disorders (confirmed by MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder.
5. Subject has suicidal ideation with intent to act within 6 months prior to screening visit or Study Day 1 (predose) based on investigator's discretion or C-SSRS, or has a history of suicidal behavior within the past year as assessed on the C-SSRS; or subject has homicidal ideation/intent at screening visit or on Day 1.
6. Subject had previously no treatment response to ketamine, S-ketamine, R-ketamine, all of the available AD treatment options in the double-blind phase (based on MGH-ATRQ), or an adequate course of electroconvulsive therapy (defined as at least 7 treatments with unilateral/bilateral electroconvulsive therapy [ECT]), in the current major depressive episode according to clinical judgment.
7. Subject has a score of ≥ 5 on the STOP-Bang questionnaire, in which case obstructive sleep apnea must be ruled out (e.g., apnea-hypopnea index [AHI] must be < 30). A subject with obstructive sleep apnea can be included if he or she is using a positive airway pressure device or other treatment/therapy that is effectively treating (i.e., AHI < 30) his or her sleep apnea.
8. Subjects who meet DSM-5 criteria for moderate or severe substance or alcohol use disorder, except for nicotine or caffeine, within 6 months prior to screening visit.
9. Subjects with lifetime history of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3,4-methylenedioxymethamphetamine (MDMA) hallucinogen-related disorder are exclusionary.
10. Subjects with positive urine drug test result(s) at screening visit or predose on Day 1 for barbiturates, methadone, opiates, cocaine, phencyclidine (PCP), and amphetamine/methamphetamines will be excluded. A positive test result for cannabinoids predose on Day 1 is exclusionary.
11. Subjects with positive alcohol breath test result at screening visit or predose on Day 1, or predose on Day 8.
12. Subject has a history of malignancy within the 5 years prior to screening.
13. Subject has known allergies, hypersensitivity, intolerance, or contraindication to ketamine, S-ketamine, R-ketamine, or excipients in the investigational drug.
14. Subject has taken any prohibited therapies.
15. Subjects have received an investigational drug, treatment of ketamine, S-ketamine, R-ketamine, vaccine, or used an invasive investigational medical device within 60 days before planned Study Day 1 or currently enrolled in an investigational study.
16. Subjects are pregnant or lactating at screening visit or prior to the SC administration on Day 1 or planning to become pregnant during the study.
17. Subject has any condition or situation/circumstance for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
18. Subject has had major surgery, (e.g., requiring general anesthesia) within 2 weeks before screening visit, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
19. Subjects is an employee of the investigator or the trial site, with direct involvement in the proposed trial or other trials under the direction of the investigator or trial site, or is a family member of an employee or of the investigator.
20. Subject has a history of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HIV, HBsAg, or anti-HCV at screening visit.
21. Subject has CS ECG abnormalities at screening or predose on Day 1.
22. Subject has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression.
23. Subject has a current or past history of seizures (uncomplicated childhood febrile seizures with no sequelae are not exclusionary).
24. Subject is taking a total daily dose of benzodiazepines greater than the equivalent of 6 mg/day of lorazepam at the start of the screening phase.
25. Subjects with any underlying medical conditions where elevation of blood pressure may pose a risk (including severe cardiovascular disease, recent cerebral injury, increased intracranial pressure, intracranial bleeding, or acute stroke, unstable heart failure, untreated glaucoma) are excluded.
26. Subjects have a current or history of significant pulmonary insufficiency/condition or with a peripheral blood oxygen saturation (SpO2) of < 93% at screening visit or prior to the SC administration on Day 1.
27. Subject has uncontrolled diabetes mellitus, as evidenced by HbA1c > 9% at screening visit or history in the prior 3 months prior to screening of diabetic ketoacidosis, hyperglycemic coma, or severe hypoglycemia with loss of consciousness.
28. Subjects have a history of interstitial cystitis or bladder inflammation.
29. Subject has any factors that might increase the risk of an injection site reaction progressing to subcutaneous necrosis under the investigator's discretion (e.g., immunocompromised patients, subjects have a history of severe skin disorder or injection site reaction at abdomen, or the subject whose abdominal area is unsuitable for SC injections (e.g., nodules, lesions, excessive pigment, infected, scarring)).
30. Significant symptoms, medical conditions, or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the trial or obtaining informed consent, or may prevent the subject from safely participating in trial.
31. Subjects receiving psychotherapy of any type that began, or was changed in frequency or focus, less than 3 months before the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AEs) | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
Incidence of abnormal orthostatic blood pressure | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
Incidence of abnormal heart rate | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  Heart rate is measured as pulse
Incidence of abnormal blood oxygen saturation (pulse oximetry) | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  Pulse oximetry will be monitored continuously for 24 hours post injection to assess for any signs/symptoms of respiratory depression.
Incidence of abnormal respiratory rate | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
Incidence of abnormal body temperature | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
Incidence of abnormal 12-lead electrocardiogram (ECG) parameters | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  Subjects should rest in a supine position for at least 5 minutes before ECG collection and should refrain from talking or moving arms or legs. ECG parameters including PR interval, QRS interval, QT interval, QTc interval, QTcF interval, RR interval will be assessed.
Incidence of abnormal hematologic findings | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  Hemoglobin, hematocrit, platelet count, red blood cell (RBC) count, and white Blood Cell (WBC) count by hematologic examination
Incidence of abnormal serum chemistry test result | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  Serum levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), calcium, creatinine, chloride, creatine phosphokinase (CPK), gamma-glutamyl transferase (GGT), glucose (non-fasting), phosphate, potassium, sodium, total bilirubin, total cholesterol, total protein, bicarbonate, albumin will be assessed.
Incidence of abnormal urine test result | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  The appearance, pH, and specific gravity of urine, and the amount/presence of protein, glucose, ketones, bilirubin, blood, nitrites, leukocytes, urobilinogen, red blood cells, white blood cells, epithelia cells, crytals, casts, and bacteria will be assessed.
Incidence of abnormal urine cytologic findings | Baseline (prior to dosing) and the End of Study (Day 36) visit
  Urine cytology is a test to examine if the subject's urine contains abnormal cells. The subject will collect their urine samples once a day in sterile containers at clinical site for 3 consecutive days while screening (baseline) and at the end of study.
Incidence and severity of dissociative symptoms assessed by Clinician Administered Dissociative States Scale (CADSS) | Baseline (prior to dosing) through the End of Study (Day 36)
  CADSS is a questionnaire designed to assess dissociative symptoms. CADSS consists of 23 questions with 5-points scale, where 0 = not at all and 4 = extremely. Higher scores represent a more severe condition.
Incidence and severity of treatment-emergent sedation assessed by Modified Observer's Assessment of Alertness/ Sedation (MOAA/S) | Baseline (prior to dosing) through the End of Study (Day 36)
  MOAA/S is a 6-point ordinal scale used to measure treatment-emergent sedation. The scores range from 0 (no response to painful stimulus) to 5 (response readily to name spoken in normal tone).
Incidence and severity of potential withdrawal symptoms assessed by Physician Withdrawal Checklist; 20-item (PWC-20) | Two weeks after last investigational product administration and through the End of Study (Day 36)/Early termination or Follow up visit
  PWC-20 is a 20-item simple and accurate method to assess potential withdrawal symptoms following cessation of IP treatment. PWC-20 consists of 20 questions with 4-points scale, where 0 = not present and 4 = severe. Higher scores represent a more severe condition.
Incidence and severity of suicide ideation assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline (prior to dosing) and through the End of Study (Day 36)/Early termination or Follow up visit
  C-SSRS is a self-report suicidal ideation rating scale. The scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future. C-SSRS involes suicide ideation, intensity of ideation, suicidal behavior, and actual attempts.
Incidence and severity of four-item positive symptom subscale of the Brief Psychiatric Rating Scale (BPRS+) | Baseline (prior to dosing) and through the End of Study (Day 36)/Early termination
  The Brief Psychiatric Rating Scale (BPRS) is an 18-item rating scale which is used to assess potential treatment-emergent psychotic symptoms. The scores range from 0 (not assessed) to 7 (extremely severe). The higher score represents a worse outcome. Only the four-item positive symptom subscale (BPRS+) will be used in the study to assess treatment-emergent psychotic symptoms. BPRS+ consists of suspiciousness, hallucinations, unusual thought content, and conceptual disorganization.
Injection site tolerability based on injection site grading scale | At the time of injection and through the End of Study (Day 36)/Early termination or Follow up visit
  Injection site grading scale consists of 5 items including assessment on pain, tenderness, induration, erythema/redness, and swelling. Each item will be scaled from Grade 0 (None) to Grade 4 (potentially life threatening). The evaluation will be performed by the investigator or trained designee who will be a qualified healthcare professional.
Injection site tolerability based on injection site pain visual analog scale (VAS) | At the time of injection and through the End of Study (Day 36)/Early termination or Follow up visit
  Injection site pain will be assessed by the subject with a 100 mm VAS scale ranging from 0 to 100, where 0 represents "no pain" and 100 represents "maximum pain". The evaluation will be performed by the investigator or trained designee who will be a qualified healthcare professional.
Injection site tolerability based on injection site evaluation for potential reactions and evidence of removal | At the time of injection and through the End of Study (Day 36)/Early termination or Follow up visit
  The local injection site will be evaluated for potential reactions and evidence of removal. The evaluation will be performed by the investigator or trained designee who will be a qualified healthcare professional.

SECONDARY OUTCOMES:
Cmax for each dosing | Up to 28 days post last dose
  Maximum observed plasma concentration following administration
Tmax for each dosing | Up to 28 days post last dose
  Time to reach the maximum observed plasma concentration following administration
AUCs for each dosing | Up to 28 days post last dosing
  The AUCs is the area under the plasma concentration-time curve from time 0 to the specified time points post-dose.
t1/2 | Up to 28 days post last dosing
  Elimination half-life

OTHER OUTCOMES:
Change from baseline in Montgomery Asberg Depression Rating Scale (MADRS) total score | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each scored from 0 (symptoms not present or normal) to 6 (severe or continuous presence of symptoms). Total score is 60. The higher MADRS total score, the more severe depression.
Clinical Global Impression - Severity (CGI-S) | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  The CGI-S provides measure of severity of subject's mental illness at the time of assessment. CGI-S is scored from 0 to 7. Considering total clinical experience, subject is assessed on severity of mental illness according to: 0 = not assessed; 1 = normal (not at all ill); 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill.
Clinical Global Impression - Improvement (CGI-I) | Since 2 hours post injection through the End of Study (Day 36)/Early termination or Follow up visit
  The CGI-I is designed to assess how much the subject's mental illness has improved or worsened relative to a baseline state at the beginning of the intervention. CGI-I is scored from 0 to 7. Subjects is assessed according to: 0 = not assessed; 1 = very much improved since the initiation of treatment; 2 = much improved; 3 = minimally improved; 4 = no change from baseline (the initiation of treatment); 5 = minimally worse; 6 = much worse; 7 = very much worse since the initiation of treatment.
Generalized Anxiety Disorder 7-item Scale (GAD-7) | Baseline (prior to dosing) through the End of Study (Day 36)/Early termination or Follow up visit
  GAD-7 is a brief and validated 7-item self-report assessment of overall anxiety. Subject responds to each item using a 4-point scale with response categories of 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety.
Response, defined as a ≥ 50% reduction from baseline in MADRS total score | Since 2 hours post injection through the End of Study (Day 36)/Early termination or Follow up visit
Remission, defined as a MADRS total score ≤ 10 | Since 2 hours post injection through the End of Study (Day 36)/Early termination or Follow up visit

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pillar Clinical Research, Little Rock, Arkansas
  - Arch Clinical Trials, St Louis, Missouri
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio